CLINICAL TRIAL: NCT01227681
Title: A Double-Blind, Placebo-Control, Study of the Neuro-protective Effect of Granulocyte-colony Stimulating Factor on Early Stage Parkinson's Disease
Brief Title: Study of the Neuro-protective Effect of Granulocyte-colony Stimulating Factor on Early Stage Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in Recruitment
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCSP-01
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- high dose G-CSF (Experimental): high dose group: 3.3ug/kg/day for consecutive 5 days of each 60 day cycle (6 cycles)
  Interventions: Drug: G-CSF
- low dose G-CSF (Active Comparator): low dose group: 1.65ug/kg/day for consecutive 5 days of each 60 day cycle (6 cycles)
  Interventions: Drug: G-CSF
- placebo (Placebo Comparator): Sodium Chloride (NaCl) 0.9 %
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: G-CSF — G-CSF(granulocyte-colony stimulating factor) is planned injected subcutaneously
  Other Names: Filgrastim, Kirin, Japan
  Arms: high dose G-CSF; low dose G-CSF
Drug: Placebo — Sodium Chloride (NaCl) 0.9 %
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of neuroprotection from granulocyte colony-stimulating factor on Parkinson disease

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease and the severity of PD still progress during the ensuing years. Currently, there is no promising medical or surgical treatment to abrogate the disease deterioration. Granulocyte colony-stimulating factor (G-CSF), one of hematopoietic growth factors, has been routinely used for hematologic disorders and stem cell harvest from normal subject. G-CSF also demonstrated neuroprotection for rodents PD model. We hypothesize G-CSF will exert the effectiveness of neuroprotection for PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn & Yahr stage I~III
* Patients with idiopathic Parkinson's disease(PD), who meet the United Kingdom Parkinson's Disease Society Brain Bank diagnostic criteria, with a good response to levodopa
* The onset of PD symptoms must be occurred > = 40 years of age (to exclude YOPD), and the patient must have been diagnosed with idiopathic PD > =40 years of age
* Patients may have symptoms of wearing OFF and/or levodopa induced dyskinesia
* Patients must rate between Hoehn & Yahr stage I to III, when in an OFF medication state
* Patients must in their optimal medication treatment state, and will not changing their medications within 3 months before and after enrollment

Exclusion Criteria:

* Patients who are proved to be Young Onset Parkinson's Disease (YOPD) and/or genetically related (e.g. Parkin).
* Women of child-bearing potential, pregnant or lactating.
* Patients who are proved to have tumor growth and/or malignancy.
* Patients with a past (within one year) or present history of psychotic symptoms requiring anti- psychotic treatment.
* Patients with active symptoms of major depression with suicidal ideation or suicide attempt.
* Patients with previous brain surgery (including pallidotomy and deep brain stimulation).
* Patients with significant cognitive impairment ( Mini-Mental State Examination, MMSE < 24).
* Patients who do not sign the inform consent,

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shin Yuan Chen, MD, Principal Investigator — Buddhist Tzu Chi General Hospital, Hualien
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parkinson's disease research center, Tzu Chi Hospital
Pre-assignment Details: No participants were randomized to receive 1.65ug/kg/day of G-CSF and placebo
Groups:
- G-CSF: 3.3ug/kg/day for consecutive 5 days of each 60 day cycle
- Low Dose G-CSF: 1.65ug/kg/day for consecutive 5 days of each 60 day cycle
- Placebo: subcutaneous Normal saline for consecutive 5 days of each 60 day cycle
Period: Overall Study
Arm/Group | G-CSF | Low Dose G-CSF | Placebo
Started | 4 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Dose G-CSF Injection for Parkinson's Disease: 3.3 ug/kg/day for consecutive 5 days of each 60 day cycle
- Low Dose G-CSF Injection for Parkinson's Disease: 1.65 ug/kg/day for consecutive 5 days of each 60 day cycle
- Placebo: normal saline 0.9% injection
- Total: Total of all reporting groups
Arm/Group | High Dose G-CSF Injection for Parkinson's Disease | Low Dose G-CSF Injection for Parkinson's Disease | Placebo | Total
Number analyzed (Participants) | 4 | 0 | 0 | 4
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 4 |  |  | 4
  >=65 years | 0 |  |  | 0
Age, Continuous [Mean (Full Range); unit: years] | 49.25 [42 to 56] |  |  | 49.25 [42 to 56]
Gender [Number; unit: participants]
  Female | 0 |  |  | 0
  Male | 4 |  |  | 4
Region of Enrollment [Number; unit: participants]
  Taiwan | 4 |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Motor Performance of Unified Parkinson's Disease Rating Scale
Description: To assess Unified Parkinson's Disease Rating Scale part III (motor function) scores from baseline Medication-off status to Medication-off status after G-CSF injection one year. Scores of UPDRS Part III ranges from 0 to 108 and higher values indicate worse outcome.
Time Frame: 2 years
Measure: Mean (Full Range); unit: scores on a scale
Groups:
- G-CSF Injection for Parkinson's Disease: 3.3ug/kg/day for consecutive 5 days of each 60 day cycle
Arm/Group | G-CSF Injection for Parkinson's Disease
Number analyzed (Participants) | 4
scores on a scale
  Baseline | 23 [17 to 27]
  post G-CSF one year | 22 [18 to 25]
Statistical Analysis 1: Comparison: G-CSF Injection for Parkinson's Disease; Null hypothesis: there is significant deterioration of UPDRS part III scores from baseline to post G-CSF injection one year; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | G-CSF Injection for Parkinson's Disease
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF Injection for Parkinson's Disease (N=4)
Musculo-skeletal soreness (Musculoskeletal and connective tissue disorders) | 3 — 3/4 participants had soreness during 5 days G-CSF injection period and discomfort can be mitigated by NSAID or Acetaminophen

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes